CLINICAL TRIAL: NCT03145142
Title: PREMOD2 NIRS Substudy - A Randomized Trial of Cerebral Oxygen Saturation in Infants Randomized to Umbilical Cord Milking or Delayed Cord Clamping
Brief Title: PREMOD2 With Near Infrared Spectroscopy Sub-study
Acronym: PREMOD2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sharp HealthCare (Other)
Collaborators: University of Ulm (Other); University College Cork (Other); University of Alberta (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREMOD2 - NIRS Sub-study; 1R01HD088646-01A1 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Hypoxia, Brain; Premature Birth
Keywords: Near-Infrared Spectroscopy
MeSH Terms: conditions — Hypoxia, Brain; Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): Milking the umbilical cord 4 times towards the infant at a speed of 20cm over 2 seconds.
  Interventions: Procedure: Umbilical cord milking
- Delayed Cord Clamping (Active Comparator): Delayed clamping of the umbilical cord for at least 60 seconds.
  Interventions: Procedure: Delayed Cord Clamping

INTERVENTIONS:
Procedure: Umbilical cord milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before it is clamped. The procedure infuses a placental transfusion of blood into the preterm infant and can be done in 15-20 seconds
  Arms: Umbilical Cord Milking
Procedure: Delayed Cord Clamping — At delivery, delayed cord clamping will be performed by having the delivering obstetrician delay clamping of the umbilical cord for at least 60 seconds.
  Arms: Delayed Cord Clamping

SUMMARY:
Early hemodynamic effects (within 3 hours of life) of Delayed Cord Clamping compared to Umbilical Cord Milking are still unknown. Four sites experienced in the use of NIRS and who have appropriate data collection equipment in the delivery room (Alberta, Ulm, Cork and San Diego) will obtain and report the physiological changes with UCM and DCC from birth until 24 hours of life. This data will yield the largest available sample of continuously recorded heart rate, cerebral tissue oxygenation, peripheral oxygen saturation, airway pressure, and administered FiO2 to delineate the short term responses to two methods of placental transfusion. In our initial trial we demonstrated increased blood pressure from 3-15 HOL with UCM compared to DCC in premature newborns <32 weeks, but did not show any differences in cerebral oxygenation.

DETAILED DESCRIPTION:
This substudy will include 400 infants <28 weeks GA enrolled in the PREMOD2 trial. Once the newborn has been delivered, received the intervention (UCM or DCC), and been placed on the resuscitation bed a NIRS sensor and a pulse oximeter will be placed within 60 seconds. While arterial saturation and heart rate data will be available to the clinical team, data from NIRS will be blinded. Data on all study infants will be recorded for at least the first 10 minutes in the delivery room, and then for 24 hours in the NICU. Heart rate, oxygen saturations, and cerebral oxygenation, will be downloaded as per each site's practice for neonatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* 23 weeks 0 days to 27 weeks 6 days.
* Enrolled in PREMOD2 trial.

Exclusion Criteria:

* NIRS Device not available
* Research Personnel not available

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
StO2 - 10M | 1st 10 minutes of life
  Cerebral Tissue Oxygen Saturation in the Delivery Room

SECONDARY OUTCOMES:
StO2 - 24H | 1st 24 hours of life
  Cerebral Tissue Oxygen Saturation in the NICU
HR - 10M | 1st 10 minutes of life
  Heart Rate in the Delivery Room
HR 24H | 1st 24 hours of life
  Heart rate in the NICU
Blood Pressure NICU | 2st 24 hours of life
  Mean Blood Pressure in the 1st 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Anup C Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns
Locations (4):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States
- Governors of University of Alberta, Edmonton, Alberta, Canada
- University of ULM, Ulm, Baden-Wurttemberg, Germany
- Cork University Maternity Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katheria AC, Szychowski JM, Essers J, Mendler MR, Dempsey EM, Schmolzer GM, Arnell K, Rich WD, Hassen K, Allman P, Varner M, Cutter GR, Finer N. Early Cardiac and Cerebral Hemodynamics with Umbilical Cord Milking Compared with Delayed Cord Clamping in Infants Born Preterm. J Pediatr. 2020 Aug;223:51-56.e1. doi: 10.1016/j.jpeds.2020.04.010. Epub 2020 May 29. PMID 32482392
- See also: PREMOD2 main trial — https://clinicaltrials.gov/show/NCT03019367